CLINICAL TRIAL: NCT01614860
Title: Identification of Patient Phenotypes Associated With Elevated Aldosterone Levels
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Peter Pang, Associate Professor of Emergency Medicine, Northwestern University
Other Study IDs: KL2-2012NWAHF; KL2RR025740 (NIH)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Acute Heart Failure
Keywords: Aldosterone; Echocardiography; Neurohormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma storage for potential future studies with existing or novel biomarkers.
Oversight: Data Monitoring Committee: No

SUMMARY:
Post-discharge mortality and re-hospitalization for acute heart failure (AHF) affects 15% and 30% of patients respectively, within 90 days. With over 1 million annual hospitalizations and a financial cost exceeding 20 billion dollars, AHF is a major public health burden. Yet no AHF therapy to date definitively reduces morbidity and mortality, and in stark contrast to heart attack patients, highly rated evidence in guidelines do not exist. Although AHF is a syndrome and not one disease, typical treatment of patients hospitalized with AHF suggests otherwise. Despite substantial differences among AHF patients, therapy is largely uniform; patients receive medicine to help get rid of excess volume and little else. Although decades of empirical use support the symptomatic benefits of traditional therapies, outcomes remain extremely poor. As opposed to the "one-size-fits-all" approach used unsuccessfully to date in clinical trials, identification of specific AHF patient sub-groups is critical, so that tailored therapies can be developed and tested. Preliminary data suggests that the neurohormone aldosterone may be detrimental in AHF patients. Furthermore, this hormone level appears to rise during hospitalization. The investigators therefore propose to identify specific AHF patient phenotypes associated with high serum aldosterone levels to subsequently address the hypothesis that early aldosterone blockade continued throughout hospitalization will decrease re-hospitalization and mortality. Specifically, the investigators hypothesize that AHF patients with elevated serum aldosterone levels have a distinct phenotype compared to those with lower or normal aldosterone levels. Specifically, they will be older, have a lower systolic blood pressure, lower EF, worse renal function, higher BNP, and previous hospitalization for HF.

ELIGIBILITY:
Inclusion criteria:

* Male or female ≥ 18 years of age
* AHF is the primary working diagnosis for ER management and treatment Have received or will receive IV diuretic therapy
* Enrolled within 12 hours of initial diuretic dose order

Exclusion criteria:

* Serum Cr ≥ 2.5mg/dL (males) or 2.0mg/dL (females), or eGFR < 20 ml/min/1.73m2
* Serum potassium ≥ 5.5 mEq/L
* Transplant recipients of any kind
* Fever > 101.0
* Severe lung disease (required home O2 or daily oral steroids)
* Acute coronary syndrome within last 30 days
* Major surgery within last 30 days
* Known hypertrophic obstructive cardiomyopathy, pericardial constriction, or hemodynamically significant valvular disease
* Life expectancy less than 12 months for any reason
* Current treatment for any malignancy of any kind
* Cardiogenic shock and/or requiring IV inotropic therapy
* Pregnant or recently pregnant within last 90 days
* Known intolerance to aldosterone antagonist
* Inability to give appropriate written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the Emergency Department (ED) with signs and symptoms of AHF
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
There is no prespecified primary outcome as this is an exploratory study | 2 years

SECONDARY OUTCOMES:
There is no secondary outcome as this is an exploratory study | 2 years

OTHER OUTCOMES:
To prospectively examine the baseline and dynamic phenotype of AHFS patients in relation to aldosterone levels on initial presentation. | two years
  Hypothesis 2.1: The "high aldosterone" phenotypic profile identified in Aim 1 will be associated with high aldosterone levels on initial presentation to the ER in our prospective replication study.
  Hypothesis 2.2: AHFS patients with high aldosterone levels on presentation will have increased high-sensitivity troponin release and echocardiographic markers of increased myocardial and atrial fibrosis.
  Hypothesis 2.3: Repeat examination at 48 hours after initial presentation will demonstrate lack of improvement in laboratory and echocardiographic biomarkers of congestion, myocyte injury, and fibrosis in AHFS patients with high aldosterone levels, suggesting a time-sensitive component to aldosterone antagonism in AHFS.

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Pang, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States